CLINICAL TRIAL: NCT02938598
Title: Optimizing a Pediatric Intervention to Increase Maternal Depression Care-Seeking
Brief Title: Motivating Our Mothers 2
Acronym: MOM2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: 800492; K23MH101157 (NIH)
Record Dates: First submitted 2016-10-17; First posted 2016-10-19 (Estimated); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Depression; Maternal Care Patterns
Keywords: maternal depression; pediatric-based maternal depression screening; maternal health services
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- A (Experimental): Engagement On - Problem Solving High - Motivation On
  Interventions: Behavioral: Maternal Depression Education and Care-Seeking Motivation
- B (Experimental): Engagement On - Problem Solving Low - Motivation On
  Interventions: Behavioral: Maternal Depression Education and Care-Seeking Motivation
- C (Experimental): Engagement On - Problem Solving High - Motivation Off
  Interventions: Behavioral: Maternal Depression Education and Care-Seeking Motivation
- D (Experimental): Engagement On - Problem Solving Low - Motivation Off
  Interventions: Behavioral: Maternal Depression Education and Care-Seeking Motivation
- E (Experimental): Engagement Off - Problem Solving High - Motivation On
  Interventions: Behavioral: Maternal Depression Education and Care-Seeking Motivation
- F (Experimental): Engagement Off - Problem Solving Low - Motivation On
  Interventions: Behavioral: Maternal Depression Education and Care-Seeking Motivation
- G (Experimental): Engagement Off - Problem Solving High - Motivation Off
  Interventions: Behavioral: Maternal Depression Education and Care-Seeking Motivation
- H (Experimental): Engagement Off - Problem Solving Low - Motivation Off
  Interventions: Behavioral: Maternal Depression Education and Care-Seeking Motivation

INTERVENTIONS:
Behavioral: Maternal Depression Education and Care-Seeking Motivation — Multicomponent behavioral and educational intervention. The investigators are only testing 3 components: Engagement, Problem-Solving, and Follow-Up Motivation

SUMMARY:
Mothers with symptoms suggesting clinical depression can be identified and potentially motivated to seek further care during pediatric visits for their young children. The best ways for pediatric providers to encourage mothers to seek further evaluation and treatment for their depressive symptoms are not known. The investigators plan to provisionally optimize a pediatric office-based intervention that the investigators developed to motivate mothers who may be depressed to seek further care and, thereby to improve the well-being of women from diverse backgrounds and their children.

DETAILED DESCRIPTION:
Depression in mothers parenting young children is common and undertreated. Depression is debilitating for mothers, negatively affects their parenting, and is associated with mental, behavioral, and physical health problems in their children. Identifying and treating mothers with depression improves both the mothers' well-being and their children's mental and overall health. Pediatric visits offer a potential significant opportunity to intervene. Mothers may see their child's pediatric provider more often than their own, and these providers could motivate mothers to seek effective, underutilized, formal depression care, by communicating how recovery from depression is linked to child well-being.

Therefore, in recent pilot work, the investigators developed a pediatric setting-based intervention that includes a validated maternal depression screen, and subsequent depression education and care-seeking motivational messages that emphasize the benefits of maternal depression care for children. Initial testing demonstrated that depression screen-positive mothers receiving the intervention had greater intention and attempts to seek depression care compared to mothers receiving usual care. The investigators then professionally translated the intervention into Spanish as a first step in increasing the generalizability of the intervention through refinement in future studies. As is often the case with interventions tested as a package, the investigators lack empirical evidence on which components of the pilot intervention deliver the greatest effects. Therefore, the investigators propose to adopt a rapid-cycle intervention improvement approach.

In this trial, the investigators will assess the effects intervention refinements on depression screen-positive mothers' depression care-seeking, using a factorial randomized design. The resulting intervention will be provisionally optimized by including only those refined components found to be most experimentally efficacious. This provisionally optimized intervention will have a higher probability of demonstrating reproducible effectiveness, potentially speeding the way to implementation. The ultimate optimized intervention will improve maternal depression care by being an essential link in future integrated systems between pediatric-based maternal depression screening and effective community-based programs for maternal mental health care.

The investigators modified the initial anticipated sample size reported from 312 to 80. During the course of recruiting and enrollment investigators found the need to reorient the trial to one of feasibility and reduced the sample size accordingly. The investigators' goal is to obtain an analytic sample size that will allow for balanced numbers of participants in each cell across sites, with a minimum of 5 observations per intervention type. Given variable recruiting and retention rates, this could be a recruited sample size between 48 and 80 individuals. In addition, investigators extended the initial recruiting time frame.

ELIGIBILITY:
Inclusion Criteria:

* primarily responsible for the day-to-day care of and obtaining pediatric care for the child with which they are presenting to the pediatric clinic;
* speak and read English or Spanish well enough to participate effectively in guided discussion;
* positive maternal depression screen;
* child aged 0-12 years;
* presenting only for well-child care;
* not currently under active and regular care for depression;
* not previously enrolled in the study.

Exclusion Criteria:

- unable to consent

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-10; Primary Completion 2019-05-23 (Actual); Study Completion 2019-05-23 (Actual)

PRIMARY OUTCOMES:
Attempt to Contact a Maternal Depression Resource | 2 Weeks Post-Intervention

SECONDARY OUTCOMES:
Intention to Contact a Maternal Depression Resource | 2 Weeks Post-Intervention

CONTACTS AND LOCATIONS:
Overall Officials: Erik O Fernandez y Garcia, MD MPH, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis, Department of Pediatrics, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2017-08-14): https://cdn.clinicaltrials.gov/large-docs/98/NCT02938598/ICF_000.pdf